CLINICAL TRIAL: NCT02246959
Title: Comparative Effectiveness of Process and Outcomes Incentives for Lipid Management
Brief Title: Process Versus Outcomes Incentives for Lipid Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Rutgers University (Other); University of California, San Francisco (Other); Carnegie Mellon University (Other); Lancaster General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL118195-01A1 (NIH)
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diabetes; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: In a 4-arm, randomized controlled trial, we propose to evaluate the relative effectiveness and cost-effectiveness of improving cholesterol levels among participants who are at high risk of CVD and who have elevated LDL cholesterol levels by testing process versus outcomes financial incentives. Participants will use electronic pill bottles that continuously monitor statin adherence.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control Arm (No Intervention): Arm 1 will be the Control arm, in which participants receive electronic pill bottles for their statin medication but are not enrolled in the sweepstakes.
- Process Arm (Experimental): Arm 2 will be a Process incentive arm where participants receive electronic pill bottles for their statin medication. In addition, this group is enrolled in a sweepstakes, in which participants may win money if they remember to take their medication.
  Interventions: Behavioral: Process Incentive
- Outcome Arm (Experimental): Arm 3 will be an Outcome incentive arm where participants receive electronic pill bottles for their statin medication. In addition, this group may receive incentives if they lower their LDL.
  Interventions: Behavioral: Outcome Incentive
- Process Plus Outcome Arm (Experimental): Arm 4 will be a process plus outcome incentive arm where participants receive electronic pill bottles for their statin medication. In addition, this group is enrolled in a sweepstakes, in which participants may win money if they remember to take their medication and receive additional incentives for lowering their LDL cholesterol.
  Interventions: Behavioral: Process Incentive; Behavioral: Outcome Incentive

INTERVENTIONS:
Behavioral: Process Incentive — Daily sweepstake conditional on daily medication adherence
  Arms: Process Arm; Process Plus Outcome Arm
Behavioral: Outcome Incentive — Incentives conditional on LDL cholesterol reduction
  Arms: Outcome Arm; Process Plus Outcome Arm

SUMMARY:
In a 4-arm, randomized controlled trial, we will evaluate the relative effectiveness and cost-effectiveness of improving cholesterol levels among participants who are at high risk of CVD and who have elevated LDL cholesterol levels by testing process versus outcomes financial incentives. Participants will use electronic pill bottles that continuously monitor statin adherence. The primary outcome will be change in LDL cholesterol over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at high risk of a cardiac event, specifically one of the following:
* Individuals with clinical ASCVD (defined as diagnosis with myocardial infarction, stroke, or peripheral vascular disease) with an LDL greater than or equal to 100 mg/dl ;
* Individuals with Diabetes (between the ages of 40-75) with an LDL greater than or equal to 100 mg/dl;
* Individuals without clinical ASCVD or diabetes with LDLC with an LDL greater than or equal to 100 mg/dl and estimated 10-year ASCVD risk 7.5%;
* Individuals without clinical ASCVD or diabetes with LDL cholesterol 190 mg/dl
* A prescription filled for a statin medication within the last 12 months (derived from pharmacy records);
* Low medication adherence on self-report completed during enrollment

Exclusion Criteria:

* Under 18 years old
* A contraindication to further statin use or have suffered statin side effects, such as myopathy
* Will not or cannot give consent
* A history of active or progressive liver disease
* Participating in another clinical trial with related aims
* Co-morbidities likely to lead to death within a short period (e.g. metastatic cancer)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2015-02; Primary Completion 2018-05 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in LDL cholesterol from baseline to 12 months | 12 months

SECONDARY OUTCOMES:
Statin Adherence | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; Peter Reese, MD, MSCE, Principal Investigator — University of Pennsylvania; Iwan Barankay, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Reese PP, Barankay I, Putt M, Russell LB, Yan J, Zhu J, Huang Q, Loewenstein G, Andersen R, Testa H, Mussell AS, Pagnotti D, Wesby LE, Hoffer K, Volpp KG. Effect of Financial Incentives for Process, Outcomes, or Both on Cholesterol Level Change: A Randomized Clinical Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2121908. doi: 10.1001/jamanetworkopen.2021.21908. PMID 34605920
- [Derived] Russell LB, Norton LA, Pagnotti D, Sevinc C, Anderson S, Finnerty Bigelow D, Iannotte LG, Josephs M, McGilloway R, Barankay I, Putt ME, Reese PP, Asch DA, Goldberg LR, Mehta SJ, Tanna MS, Troxel AB, Volpp KG. Using Clinical Trial Data to Estimate the Costs of Behavioral Interventions for Potential Adopters: A Guide for Trialists. Med Decis Making. 2021 Jan;41(1):9-20. doi: 10.1177/0272989X20973160. Epub 2020 Nov 20. PMID 33218296